CLINICAL TRIAL: NCT04120129
Title: An Investigation of Transcranial Magnetic Stimulation (TMS) for Trigeminal Neuralgia (TGN)
Brief Title: Transcranial Magnetic Stimulation (TMS) for Trigeminal Neuralgia
Acronym: TGN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Mark Witcher, Neurosurgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-371
Record Dates: First submitted 2019-08-23; First posted 2019-10-09 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Facial Pain
Keywords: trigmenial neuralgia; Chronic orofacial pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Intervention Model Description: TMS, sham-TMS, and no treatment groups
Who Masked: Participant, Investigator
Masking Description: TMS and sham TMS treatment group participants and researchers will be blinded to which treatment the participant receives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TMS treatment (Experimental): participants receive TMS treatment
  Interventions: Device: TMS
- sham TMS (Sham Comparator): participants receive control TMS treatment
  Interventions: Device: sham TMS coil
- non intervention (No Intervention): control group

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation (TMS) is a noninvasive brain stimulation technique which produces short pulsatile magnetic fields (similar to that of an MRI) via two extracranial, figure 8-shaped electric coils which can induce a small, temporary, electric current in the brain currently approved and used for depression.
  Other Names: TMS coil
  Arms: TMS treatment
Device: sham TMS coil — The sham TMS does cause some stimulation to the participant so that the participants get the sensation of treatment without any cortical excitation that TMS delivers. The sensation experienced is similar to the muscle twitching or finger tapping experienced by TMS participants.
  Arms: sham TMS

SUMMARY:
The primary objective is to establish the feasibility of using TMS for COFP pain management in the interim period before surgery. This will be investigated by comparing the non-intervention group's self-reported pain to those who recieved TMS at several timepoints.

DETAILED DESCRIPTION:
Participants will be randomized to either receive transcranial magnetic stimulation (TMS), Sham-TMS (a non-therapeutic TMS coil which sounds and feels similar to normal TMS), or standard treatment during the weeks of wait time before surgery for chronic orofacial pain (COFP). TMS is a noninvasive, painless magnetic device which, when applied to the head for a few minutes, has been shown to reduce pain in people with COFP. The sham TMS is a sub-therapeutic level of magnetcic stimulation which makes the same sound as normal TMS and causes a similar tingling of the skin.

Both those who receive this new pain intervention and those who do not will be asked to fill out a short online survey about their pain at several points during the study. The survey takes about 10 minutes to fill out and each of the 5 TMS sessions last 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of classic trigeminal neuralgia or persisten idiopathic facial pain
* Considered an appropriate candidate for surgical or stereotactic intervention - microvascular decompression or stereotactic radiosurgery- ( includes factors such as overall health, chronic medication, comorbidities) and patient preference
* Between ages 18-100
* Able to participate in 5 consecutive TMS treatments
* Has at least 3 weeks between pre-op visit and scheduled date of surgery
* Able to provide consent and complete online questionnaires on their own

Exclusion Criteria:

* Multiple Sclerosis or trauma-related etiology of facial pain (i.e. secondary facial pain)
* contraindication to TMS, per device guidelines:

Metallic implant in or near head Implanted stimulator on or near head recent suicidal ideation history of epilepsy, stroke, or unexplained seizure

- Need for urgent/emergent surgical decompression.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changed Pain assessed by self reported measures: Short-form McGill Pain Questionnaire 2 (SF-MPQ-2) | 7 months
  The primary objective is to establish the effectiveness of TMS for COFP pain management in the interim period before surgery. This will be investigated by comparing the non-intervention group's self-reported pain to those who received TMS at several timepoints. Short-form McGill Pain Questionnaire 2 (SF-MPQ-2)will be used. The scale asks participants to identify their pain level across body areas and total from 0-10 (0 being none & 10 worst possible)

SECONDARY OUTCOMES:
Length of altered pain | 7 months
  A secondary objective is to establish how long the effects of TMS last. This will be done by comparing self-reported pain scores prior to TMS, after TMS and at several timepoints thereafter in those who recieved the treatment. Short-form McGill Pain Questionnaire 2 (SF-MPQ-2) will be used. The scale asks participants to identify their pain level across body areas and total from 0-10 (0 being none & 10 worst possible)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Witcher, MD, PhD, Principal Investigator — Surgeon
Locations (1):
- Institute for Orthopedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No